CLINICAL TRIAL: NCT06477926
Title: A Phase 1 Relative Bioavailability and Food Effect Study of ABBV-668 Extended-Release Formulations
Brief Title: A Study to Assess Relative Bioavailability and Food Effect of ABBV-668 Extended-Release Formulations in Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M25-176
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; ABBV-668

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- ABBV-668 Regimen A (Experimental): Participants will receive ABBV-668 Immediate Release (IR) capsules on Day 1 under fasting conditions
  Interventions: Drug: ABBV-668 IR
- ABBV-668 Regimen B (Experimental): Participants will receive ABBV-668 Extended Release (ER) tablets Formulation 1 administered on day 1 under fasting conditions
  Interventions: Drug: ABBV-668 ER
- ABBV-668 Regimen C (Experimental): Participants will receive ABBV-668 Extended Release (ER) tablets Formulation 1 administered on day 1 under fed conditions
  Interventions: Drug: ABBV-668 ER
- ABBV-668 Regimen D (Experimental): Participants will receive ABBV-668 Extended Release (ER) tablets Formulation 2 administered on day 1 under fasting conditions
  Interventions: Drug: ABBV-668 ER
- ABBV-668 Regimen E (Experimental): Participants will receive ABBV-668 Extended Release (ER) tablets Formulation 2 administered on day 1 under fed conditions
  Interventions: Drug: ABBV-668 ER
- ABBV-668 Regimen F (Experimental): Participants will receive ABBV-668 Extended Release (ER) tablets Formulation 3 administered on day 1 under fasting conditions
  Interventions: Drug: ABBV-668 ER
- ABBV-668 Regimen G (Experimental): Participants will receive ABBV-668 Extended Release (ER) tablets Formulation 3 administered on day 1 under fed conditions
  Interventions: Drug: ABBV-668 ER

INTERVENTIONS:
Drug: ABBV-668 IR — • Oral Capsule
  Arms: ABBV-668 Regimen A
Drug: ABBV-668 ER — • Oral Tablets
  Arms: ABBV-668 Regimen B; ABBV-668 Regimen C; ABBV-668 Regimen D; ABBV-668 Regimen E; ABBV-668 Regimen F; ABBV-668 Regimen G

SUMMARY:
The objectives of this study are to assess safety and tolerability of the new ABBV-668 ER tablets, to assess the oral bioavailability of the ABBV-668 ER tablets relative to the ABBV-668 IR capsules, and to assess the pharmacokinetics of the ER tablets under fasting and fed conditions in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI is ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at screening.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of any clinically significant sensitivity or allergy to any medication or food.
* History of any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* Participant using any medication, vitamins and/or herbal supplements (including traditional Chinese medicine), with the exception of hormonal replacement therapies for females, on a regular basis.
* Any use of tobacco or nicotine-containing products within 180 days prior to the first dose of study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-668 | Up to approximately 47 days
  Cmax of ABBV-668
Time to Cmax (Tmax) of ABBV-668 | Up to approximately 47 days
  Tmax of ABBV-668
Terminal Phase Elimination Rate Constant (Beta) of ABBV-668 | Up to approximately 47 days
  Terminal phase elimination rate constant (beta) of ABBV-668
Terminal Phase Elimination Half-Life (t1/2) of ABBV-668 | Up to approximately 47 days
  Terminal phase elimination half-life of ABBV-668
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-668 | Up to approximately 47 days
  AUCt of ABBV-668
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-688 | Up to approximately 47 days
  AUCinf of ABBV-688
Number of Participants With Adverse Events (AEs) | Up to Day 47
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 266960, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-176